CLINICAL TRIAL: NCT03907436
Title: The NUTRIENT Trial (NUTRitional Intervention Among myEloproliferative Neoplasms): Feasibility Phase
Acronym: NUTRIENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Angela G. Fleischman, Assistant Professor, Division of Hematology/Oncology, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-4521; 18-30 (Other: Chao Family Comprehensive Cancer Center)
Record Dates: First submitted 2019-04-02; First posted 2019-04-09 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Myeloproliferative Disorder; Myeloproliferative Syndrome; Myelofibrosis; Polycythemia Vera; Essential Thrombocythemia
Keywords: nutrition; diet; inflammation; myeloproliferative neoplasm
MeSH Terms: conditions — Myeloproliferative Disorders; Primary Myelofibrosis; Polycythemia Vera; Thrombocythemia, Essential; Inflammation | interventions — Diet, Mediterranean

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two healthy diets (USDA or Mediterranean diet)
Who Masked: Participant
Masking Description: Participants will not be told which diet arm they are randomized to. Participants will not be told the two options are USDA or Mediterranean, only there are two "healthy" diets.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- USDA diet arm (Sham Comparator): Participants will receive dietician counseling based on the USDA guidelines for Americans, 2010. Participants will receive 10 weekly pdf handouts via email with information pertaining to these diet recommendations. Participants will receive same surveys (including 14 point Mediterranean diet adherence score), 24 hour diet recalls, and biological sample draws at the Mediterranean arm.
  Interventions: Other: USDA Diet
- Mediterranean diet arm (Experimental): Participants will receive dietician counseling on a standard Mediterranean diet although they will not be told this diet is labelled as a Mediterranean diet. Participants will receive 10 weekly pdf handouts via email with information pertaining to these diet recommendations. Participants will receive same surveys (including 14 point Mediterranean diet adherence score), 24 hour diet recalls, and biological sample draws at the USDA diet arm.
  Interventions: Other: Mediterranean Diet

INTERVENTIONS:
Other: USDA Diet — Participants will receive counseling and education on USDA Guidelines for Americans, 2010
  Arms: USDA diet arm
Other: Mediterranean Diet — Participants will receive counseling and education on a Mediterranean diet.
  Arms: Mediterranean diet arm

SUMMARY:
The purpose of this study is to determine whether MPN patient are able to adhere to a dietary intervention. Participants will be randomized to one of two healthy diets. Participants will receive in person dietician counseling and online curriculum. Adherence will be measured using online surveys and phone diet recalls. Changes in inflammatory markers in blood will also be measured at 5 time points during this 15 week study.

DETAILED DESCRIPTION:
This is a 15 week study, including 10 weeks of active diet intervention. Each participant will receive one dietician counseling session at the beginning of the diet intervention period, two brief follow up dietician phone calls, and 10 diet education handouts delivered via email each week. The main objective of this protocol is to test whether MPN patients can adhere to a diet intervention. The investigators will measure adherence in both arms with patient reported diet recall every two weeks via internet surveys. As exploratory endpoints the investigators will measure changes in inflammatory markers, symptom burden, physical activity level, sleep, and gut microbiome in participants over the course of the study. If successful, the investigators plan to use this intervention in a larger trial to assess whether a diet intervention can effectively change symptom burden and inflammation in MPN patients.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Diagnosis of Myeloproliferative Neoplasm (MPN) including Essential Thrombocythemia (ET), Polycythemia Vera (PV), or Myelofibrosis (MF)
* Any type of previous therapy is allowed
* ECOG performance status ≤2
* Life expectancy of greater than 20 weeks
* Has an email address and can access the internet
* Able to read and understand English

Exclusion Criteria:

* Children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
14-point Mediterranean Diet Adherence Screener (MEDAS) | 15 weeks
  14 question survey assessing adherence to a Mediterranean diet. This is a 14 question survey, with possible 1 point per question. A perfect adherence to a Mediterranean Diet is 14 on this survey (min 0 max 14). Higher values represent closer adherence to a Mediterranean diet.

SECONDARY OUTCOMES:
Myeloproliferative Neoplasm Symptom Assessment Form Total Symptom Score (MPN-SAF TSS) | 15 weeks
  MPN Symptom Assessment Form Total Symptom Score (MPN-SAF TSS) score, a validated measure for quantifying symptom burden in MPN. This is a 10 item survey, with each question answered on a scale of 0 to 10. The minimum score is 0, the maximum score is 100. Higher numbers mean a higher symptom burden.
Inflammatory cytokines | 15 weeks
  Measurement of inflammatory cytokines in the plasma. This includes EGF, Eotaxin, FGF-basic, G-CSF, GM-CSF, HGF, IFN-alpha, IFN-gamma, IL-1 beta, IL-1 alpha, IL-1RA, IL-2, IL-2R, IL-3, IL-4, IL-5, IL-6, IL-7, IL-8, IL-9, IL-10, IL-12 (p40/p70) IL-13, IL-15, IL-17A, IL-17F, IL-22, IP-10, MCP-1, MIG, MIP-1 alpha, MIP-1 beta, RANTES, TNF-alpha, VEGF.

CONTACTS AND LOCATIONS:
Overall Officials: Angela G Fleischman, MD PhD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Avelar-Barragan J, Mendez Luque LF, Nguyen J, Nguyen H, Odegaard AO, Fleischman AG, Whiteson KL. Characterizing the microbiome of patients with myeloproliferative neoplasms during a Mediterranean diet intervention. mBio. 2023 Dec 19;14(6):e0230823. doi: 10.1128/mbio.02308-23. Epub 2023 Oct 25. PMID 37877698
- See also: website with more information on the diet and enrollment information — http://www.wearempn.org/interestedinenrolling

DOCUMENTS (1):
  • Informed Consent Form (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/36/NCT03907436/ICF_000.pdf